CLINICAL TRIAL: NCT00541697
Title: A Double-Blind, Multicenter Study to Assess the LDL-C Lowering of Combination Tablets Ezetimibe/Simvastatin (10mg/20mg) and Ezetimibe/Simvastatin (10mg/40mg) Compared to Atorvastatin 20mg in Patients With Type II Diabetes.
Brief Title: Eze/Simva Switch Study in Diabetics (0653A-807)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-807; MK0653A-807; 2007_645; NCT00093106 (obsolete NCT alias)
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ezetimibe; Simvastatin; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin / Duration of Treatment: 6 Weeks
Drug: Comparator: atorvastatin / Duration of Treatment: 6 Weeks

SUMMARY:
A study to assess the effectiveness and tolerability of MK0653A and MK0653A versus Atorvastatin in lowering LDL-C levels.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with Atorvastatin 10 mg for at least 6 weeks
* Have Type 2 Diabetes
* Weight must be stable for more than 6 weeks before entering the study

Exclusion Criteria:

* Consume more than 14 alcoholic drinks per week.
* Pregnant or lactating
* Have taken another investigation drug within 3 months of starting this study
* History of congestive heart failure, heart attack, coronary artery bypass surgery
* Uncontrolled high blood pressure
* HIV positive
* History of cancer in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2005-01-19 (Actual); Primary Completion 2005-09-28 (Actual); Study Completion 2005-10-14 (Actual)

PRIMARY OUTCOMES:
Determine the additional LDL-C lowering achieved by switching to MK0653A as compared to Atorvastatin after 6 weeks of treatment | 6 Weeks

SECONDARY OUTCOMES:
Determine the effect of MK0653A versus Atorvastatin on total cholesterol after 6 weeks of treatment | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Constance C, Westphal S, Chung N, Lund M, McCrary Sisk C, Johnson-Levonas AO, Massaad R, Allen C. Efficacy of ezetimibe/simvastatin 10/20 and 10/40 mg compared with atorvastatin 20 mg in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2007 Jul;9(4):575-84. doi: 10.1111/j.1463-1326.2007.00725.x. Epub 2007 Apr 19. PMID 17451425